CLINICAL TRIAL: NCT04814979
Title: Effects of Low-intensity Pulsed Ultrasound on Pain and Functional Disability in Patients With Lumbar Spondylolysis: A Randomized Controlled Trial
Brief Title: Effects of Low-intensity Pulsed Ultrasound on Pain and Functional Disability in Patients With Lumbar Spondylolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS-UIPT/690/2020
Record Dates: First submitted 2021-03-20; First posted 2021-03-24 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Spondylolysis
Keywords: lumbar vertebra; pain; functional disability; low-intensity pulsed ultrasound
MeSH Terms: conditions — Spondylolysis; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Low-intensity pulsed ultrasound along with routine physical therapy
  Interventions: Device: Low-intensity pulsed ultrasound (LIPUS); Other: Routine physical therapy
- Control Group (Active Comparator): Routine physical therapy alone
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Device: Low-intensity pulsed ultrasound (LIPUS) — Low-intensity pulsed ultrasound (LIPUS) consists of frequencies usually ranging from 0.75- 1.5 MHz at intensities <100mW/cm² (usually about 30mW/cm²) and usually pulsed at 1:4. The transducer head is strapped or otherwise held in place and remains stationary for treatment periods in the region of 20 minutes. Again, US medium is used for efficient sound transfer to deeper tissues. This modality was approved by the FDA in the United States in 1994 for the accelerated healing of fresh fractures and then approved by the same body in 2000 for the treatment of established non-union fractures. The studies presented to the FDA demonstrated that LIPUS had a positive effect during all three main stages of fracture healing, i.e. inflammatory, reparative and remodelling by enhancing angiogenesis, chondrogenesis and osteogenesis.
  Arms: Experimental Group
Other: Routine physical therapy — Gentle hamstrings stretching for 15 seconds 3 times a day. Flexibility of these muscle reduces stress to the lumbar region thus enhances the spino-pelvic rhythm (lumbar motion/pelvic motion). Strengthening of abdominal muscles (transversus abdominis and internal oblique). Training of these "stability" muscles in the lumbar spine provides a solid foundation for the individuals to integrate them into their functional movement patterns. Exercises focusing on these muscles have been shown to significantly decrease pain and disability in people with spondylolysis. Each exercise will be performed as 3 sets of 10 repetitions on alternate days.

SUMMARY:
Low-intensity pulsed ultrasound (LIPUS) is effective in accelerating the healing of fractures, reduction in costs to the state, reduction in the numbers of those patients who progress from out-patient care to long term care who, in the process lose their ability to perform activities of daily living and consequently their independence.

DETAILED DESCRIPTION:
Aim of this study was to determine the effects of low-intensity pulsed ultrasound on pain and functional disability in patients with lumbar spondylolysis. Thirty four (29 males & 5 females) diagnosed subjects of lumbar spondylolysis with symptomatic low back pain since four months aged between twenty to forty years were recruited. This randomized controlled trial was a part of PhD Physical Therapy project conducted at Department of Physiotherapy, University of Lahore Teaching Hospital, Lahore, Pakistan, from June 2020 to March 2021 by using non probability purposive sampling technique. Subjects were divided randomly into two equal groups (Group-A and Group-B). Lottery method was used to randomly assign patients into two groups. Numeric Pain Rating Scale (NPRS) was utilized to measure pain intensity and Oswestry Disability Index (ODI) to measure functional disability. Data was analyzed by using SPSS 21.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Diagnosed subjects of lumbar spondylolysis with symptomatic low back pain since four months
* Age: 20-40 years

Exclusion Criteria:

* Subjects with the history of neurological or autonomic deficits,
* Other fracture or bony abnormalities
* Rheumatic disease
* Other spinal problems
* Post-menopausal female
* Osteoporosis
* Osteopenia

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain on Numeric Pain Rating Scale at week 12 | Baseline and Week 12
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain with a reliability of 0.96 and validity 0.86. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.
  Change = (Week 12 Score - Baseline Score)
Change from Baseline in the Functional Disability on Oswestry Disability Index at week 12 | Baseline and Week 12
  The Oswestry Disability Index is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools with a reliability of 0.90 and validity 0.96. Scoring Instructions: For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. If all 10 sections are completed the score is calculated as follows:
  Example: 16 (total scored) 50 (total possible score) x 100 = 32%
  If one section is missed or not applicable the score is calculated:
  16 (total scored) 45 (total possible score) x 100 = 35.5% Minimum detectable change (90% confidence): 10% points (change of less than this may be attributable to error in the measurement) Change = (Week 12 Score - Baseline Score)

SECONDARY OUTCOMES:
Change from Baseline in Pain on Numeric Pain Rating Scale at week 20 | Baseline and Week 20
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain with a reliability of 0.96 and validity 0.86. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.
  Change = (Week 20 Score - Baseline Score)
Change from Baseline in the Functional Disability on Oswestry Disability Index at and week 20 | Baseline and Week 20
  The Oswestry Disability Index is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools with a reliability of 0.90 and validity 0.96. Scoring Instructions: For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. If all 10 sections are completed the score is calculated as follows:
  Example: 16 (total scored) 50 (total possible score) x 100 = 32%
  If one section is missed or not applicable the score is calculated:
  16 (total scored) 45 (total possible score) x 100 = 35.5% Minimum detectable change (90% confidence): 10% points (change of less than this may be attributable to error in the measurement) Change = (Week 20 Score - Baseline Score)

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Tanveer, PhD, Principal Investigator — University of Lahore
Locations (1):
- Institutional Review Board of Faculty of Allied Health Sciences, University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No